CLINICAL TRIAL: NCT01302821
Title: NCI 8701: A Pilot Study Utilizing C11 Alpha Methyl Tryptophan (AMT) PET Functional Imaging in Patients With Metastatic Invasive Breast Cancer Treated With 1 Methyl D Tryptophan Plus the Ad p53 DC Vaccine
Brief Title: C11 AMT Positron Emission Tomography (PET) Imaging in Patients With Metastatic Invasive Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCI 8701; MCC-16216 (Other: H. Lee Moffitt Cancer Center and Research Institute)
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: breast - male; breast - female; metastatic; invasive
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Vaccines; advexin; 1-methyltryptophan; alpha-methyltryptophan; Radioactive Tracers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy (Experimental): AMT positron emission tomography with integrated computed tomography (PET/CT)scanning in metastatic breast cancer patients to identify tumors with increased AMT uptake due to up-regulated IDO expression.
  Interventions: Biological: Adenovirus-p53 transduced dendritic cell vaccine; Drug: 1-methyl-D-tryptophan; Radiation: Carbon C 11 alpha-methyltryptophan

INTERVENTIONS:
Biological: Adenovirus-p53 transduced dendritic cell vaccine — The Ad.p53 DC vaccine will be injected intradermally (through the skin) into four separate sites. The patient's vaccine will be the same dose throughout the study.
  Other Names: Ad.p53 DC; vaccine; Advexin
Drug: 1-methyl-D-tryptophan — Each treatment cycle is comprised of 21 days. The treatment is continuous with no breaks in between cycles. Patients would not be allowed to take any tryptophan containing supplements while participating on this study.
  Other Names: NSC 721782; 1-MT
Radiation: Carbon C 11 alpha-methyltryptophan — The experimental examination for this research is the administration by a needle in a vein of Tryptophan labeled with a radioactive tracer (a substance is believed to enhance imaging for easier detection and measurement), Carbon 11, when when the patient has not eaten for five hours. A standard PET/CT scanner is then used to create images of the tracer a few minutes later.
  Other Names: radioactive tracer

SUMMARY:
The purpose of this research project is to create images of where and how the amino acid (the building blocks of proteins)Tryptophan is processed in normal and abnormal tissue in the patient's body. Tryptophan is a normal building block of proteins in the body. Sometimes in the case of cancer and other diseases, Tryptophan is processed abnormally, and possible treatments for this abnormality are of great interest because of the potential to improve cancer care.

DETAILED DESCRIPTION:
Coordinating Center: Southeast Phase 2 Consortium (SEP2C), Moffitt Cancer Center.

Research participation involves up to three experimental imaging examination visits in radiology: a baseline before the patient starts a cancer treatment, a follow-up a few days later, and a later follow up to see how the treatment may affect normal or abnormal processing of Tryptophan.

The research imaging results will be linked with other evidence of the patient's disease, but will not effect their care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on the NCI 8461/MCC 16025 study.
* Consent for participation in this companion imaging study and be able to successfully complete a minimum of two AMT PET/CT scans.

Exclusion Criteria:

* Patients must not meet any of the exclusion criteria for the NCI 8461/ MCC 16025 study.
* Not have any medical conditions prohibiting the successful completion of a minimum of two AMT PET/CT scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Estimated); Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Detected Changes in Regions of Interest (ROIs) | Average of 7 weeks
  Changes in C-11 AMT uptake and localization (measured by SUV) between baseline and approximately 4 days after initiation of treatment. The primary objective is to determine whether such changes can be detected in regions of interest (ROIs) using PET/CT imaging in patients with metastatic breast cancer enrolled in NCI 8461/ MCC16025. The SUV values in identified regions of interest (ROIs) for each patient will be compared over time between baseline and approximately 4 days after initiation of treatment, and after completion of the protocol treatment. The analysis will be largely exploratory and descriptive as the sample size and study design will likely preclude an adequate/definitive statistical conclusion of SUV values between the two time points.

SECONDARY OUTCOMES:
Number of Participants with Clinical Response | Average of 7 weeks
  Clinical responses based on Response Evaluation Criteria In Solid Tumors [RECIST] criteria, to 1-MT plus the Ad.p53 DC vaccine.
Number of Participants with Presence of IDO ImmunoHistoChemistry (IHC) Expression | Average of 7 weeks
  Presence of immuno-modulatory enzyme indoleamine 2,3-dioxygenase (IDO) IHC expression (positive vs. negative as described in NCI 8461/MCC 16025) in the assayed tumor sample.
Number of Participants with Immune Response | Average of 7 weeks
  Immune response to the vaccine (by ELISPOT criteria as described in NCI 8461/MCC 16025). The secondary endpoint immunologic response is defined as IFN-γ p53 T cell specific ELISPOT assay count measured, being ≥ 2 SDs above the baseline for a patient.
Number of Participants with Adverse Events | Average of 7 weeks
  Examine toxicity data of the protocol treatment according to Common Terminology Criteria for Adverse Events (CTCAE) V4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Soliman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute